CLINICAL TRIAL: NCT04286984
Title: Study of the Efficacy of a Patient Blood Management Program Implemented in Patients Undergoing Curative Gastric Cancer Resection
Brief Title: Implementation of a Patient Blood Management Program in Gastric Cancer Surgery
Acronym: IPAT
Status: Completed | Type: Observational
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Javier Osorio, Principal Investigator, Hospital Universitari de Bellvitge
Other Study IDs: IPAT
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Gastric Cancer; Anemia, Iron Deficiency; Surgery--Complications; Transfusion Related Complication
Keywords: Gastric Cancer; Anemia; Intravenous Iron; Patient Blood Management; Surgery
MeSH Terms: conditions — Stomach Neoplasms; Anemia, Iron-Deficiency; Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-upPBM: Patients with a diagnosis of gastric cancer before the upPBM implementation in their attending center
- Post-upPBM: Patients with a diagnosis of gastric cancer after the upPBM implementation in their attending center
  Interventions: Other: unified protocol of Patient Blood Management measure

INTERVENTIONS:
Other: unified protocol of Patient Blood Management measure — upPBM description: After performing a laboratory work-up 2 to 4 weeks before surgery, preoperative iron supplementation in case of iron deficiency anemia at least 7 days before surgery was recommended. Preoperative anemia was defined by a Hb level < 13 g/dL for both sexes. In anemic patients, iron status study was recommended and iron supplementation with intravenous iron was indicated if Hb<12g/dL and/or ferritin <300 mg/l. Intravenous iron (ferric sucrose or carboxymaltose) was administrated with the goal of recovering iron deficit, calculated using the Ganzoni formula or by the simplified strategy, only available for ferric carboxymaltose. Recommended transfusion triggers were: Hb < 9 g/dL for patients with risk factors and/or anemia symptoms; and Hb < 7 g/dL for the rest of patients in absence of active bleeding.
  Other Names: upPBM
  Groups: Post-upPBM

SUMMARY:
Retrospective evaluation on a prospective cohort of patients undergoing curative gastric cancer resection to evaluate the impact of a patient blood management (PBM) program on transfusion rate and clinical outcomes. The study aims to compare transfusion practices and clinical outcomes of patients undergoing elective gastric cancer resection before and after implementing a PBM program, which included strategies to detect and treat preoperative anemia and restrictive transfusion practice (2014-2018). Primary outcome is transfusion rate (TR). Secondary outcomes are transfusion index (TI), postoperative complications, length of stay, 30-day readmissions, and 90-day mortality. Adherence to protocol is also analyzed. Differences of variables before and after PBM program implementation are evaluated with mean comparing analysis adjusted by confounding factors.

DETAILED DESCRIPTION:
The Spanish EURopEan CanCer Audit (EURECCA) Esophagogastric Cancer Group is a surgical quality improvement project, linked to the EURECCA network in Europe. EURECCA's population-based registry prospectively collects clinical data from all public hospitals in the participating regions providing them with their outcomes benchmarked against other hospitals. Ninety variables with detailed definitions are prospectively collected from each patient by the reference surgeon at each institution. Validation of completeness and accuracy of data registration (period 2014-2017) has recently been performed revealing a completeness rate of 97% and an accuracy rate of 95% (ClinicalTrials.gov, NCT03541629, pending publication).

During a workshop of the Spanish EURECCA Esophagogastric Cancer Group in May 2014, a wide heterogeneity in perioperative transfusion policies among hospitals was detected. After several meetings, a unified protocol of PBM measures (upPBM) was agreed in February 2016. Briefly, the upPBM included strategies to address two PBM pillars: anemia detection and treatment according to the algorithm described in Figure 1; and a restrictive transfusion practice according to national guidelines for transfusion triggers. After performing a laboratory work-up 2 to 4 weeks before surgery, preoperative iron supplementation in case of iron deficiency anemia at least 7 days before surgery was recommended. Preoperative anemia was defined by a Hb level < 13 g/dL for both sexes. In anemic patients, iron status study was recommended and iron supplementation with intravenous iron was indicated if Hb<12g/dL and/or ferritin <300 mg/l. Intravenous iron (ferric sucrose or carboxymaltose) was administrated with the goal of recovering iron deficit, calculated using the Ganzoni formula or by the simplified strategy, only available for ferric carboxymaltose. Recommended transfusion triggers were: Hb < 9 g/dL for patients with risk factors and/or anemia symptoms; and Hb < 7 g/dL for the rest of patients in absence of active bleeding.

After consensus, the upPBM was introduced through specific workshops to the members of the local multidisciplinary team from all participating hospitals by the two principal investigators of this study, and approval was obtained from each Institutional Review Board. Start of application of upPBM was prospectively communicated to the principal investigator of the study by the reference surgeon in each center.

The aim of this study is to evaluate the implementation and efficacy of a PBM protocol on perioperative RBCT and postoperative outcomes for patients undergoing gastric cancer resection with curative intent.

This is a multicenter retrospective study on a prospective cohort of consecutive patients undergoing elective gastric cancer resection with curative intent between January 2014 and December 2018 in hospitals of the Spanish EURECCA project which implemented the upPBM before December 31th, 2017, to ensure a minimum 1-year follow-up. Patients are divided in 2 groups: those with a diagnosis of gastric cancer before the upPBM implementation in their attending center and those with a diagnosis afterwards.

Recorded data for each patient are age, sex, American Society of Anesthesiologists Classification (ASA class), Body Mass Index (BMI), percentage of unintended weight loss 6 months before surgery, Charlson Comorbidity Index (CCI) (categorized as 0, 1-2, and > 3), tumor location, tumoral pathological stage (8th edition, Union for International Cancer Control, UICC), neoadjuvant treatment, type of gastrectomy (distal subtotal or total), extension of lymphadenectomy according to the Japanese Gastric Cancer Association Classification (D), surgical approach (open or minimally invasive), associated multivisceral resection, Hb at diagnosis and before surgery, preoperative intravenous iron treatment, number of transfused units, moment of transfusion (pre- or perioperative), postoperative complications, hospital readmission and mortality. Transfusion Rate (TR) is defined as the percentage of patients receiving any RBCT over the total of patients. Transfusion Index (TI) is defined as the total number of RBC units transfused divided by the number of transfused patients. Both TR and TI are defined as preoperative (from the date of diagnosis of gastric cancer to the date of surgery), perioperative (from the date of surgery to the date of hospital discharge) or global (from the date of diagnosis to the date of hospital discharge). Postoperative complications were recorded the 30 first days after surgery, defined according to the Gastrectomy Complications Consensus Group (GCCG) and graded with the Clavien-Dindo (CD) classification. Readmissions are considered during the 30 first days after hospital discharge and mortality is recorded during the 90 first days after surgery. Failure-to-rescue was calculated as the proportion of patients with a severe complication (Clavien-Dindo score >IIIa) dying during the first 90 days after surgery.

Primary endpoints are global, preoperative and perioperative TR. Secondary endpoints were TI, Hb improvement after preoperative treatment with intravenous iron, overall, severe and infectious postoperative complications rates, length of stay, and mortality. Protocol compliance is evaluated with the following measures: determination of Hb > 14 days before surgery; determination of ferritin in patients with Hb < 13 g/dL; percentage of patients with Hb <12 g/dL and/or ferritin < 300 mg/l at diagnosis treated preoperatively with intravenous iron > 7 days before surgery; and percentage of patients transfused following upPBM threshold recommendations.

Data variables are described using counts and percentages, means and standard deviation or median and interquartile range (IQR) as needed. For basal patient, tumor and surgery characteristics, comparation before and after upPBM is done with a Chi2 study for discontinuous and t Student study for continuous variables, considering significant difference when p<0.05. For study outcomes, raw and adjusted differences before and after upPBM implementation are reported with a 95% confidence interval (CI95%).Variables used in the adjustment are possible confounding factors that, based on the investigator's previous experience and published data, could vary during the study period and have a potential impact on perioperative transfusion, postoperative morbidity and length of stay: age, CCI score, neoadjuvant treatment, type of gastrectomy (subtotal or total), minimally invasive surgery, lymphadenectomy extension (D), and visceral associated resection. To assess global, preoperative and intra + postoperative TR difference before and after upPBM implementation a zero-inflated negative binomial regression model is used. To assess postoperative complications, reoperation, hospital readmission (30 days) and postoperative mortality (90 days) difference before and after upPBM implementation a logistic regression model is used. Estimates are bounded by 95% confidence intervals. Statistical significance was held at 5%. All analyses are performed using R version 3.6.1.

ELIGIBILITY:
Inclusion Criteria:

- Patients undergoing elective gastric cancer resection with curative intent between January 2014 and December 2018 in hospitals of the Spanish EURECCA project which implemented the upPBM before December 31th, 2017.

Exclusion Criteria:

* Metastasis
* Palliative Surgery
* Hospitals non implementing the upPBM before December 31th, 2017

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multicenter study on a prospective cohort of consecutive patients undergoing elective gastric cancer resection with curative intent between January 2014 and December 2018 in hospitals of the Spanish EURECCA project which implemented the upPBM before December 31th, 2017, to ensure a minimum 1-year follow-up of upPBM.
Sampling Method: Non-Probability Sample
Enrollment: 1063 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Transfusion Rate | 2014-2018
  Percentage of patients receiving any red blood cell trasfusion over the total of patients

SECONDARY OUTCOMES:
Transfusion Index | 2014-2018
  Total number of red blood cell units transfused divided by the number of transfused patients
Rate of postoperative complications | 2014-2018
  Postoperative complications recorded the 30 first days after surgery, defined according to the Gastrectomy Complications Consensus Group (GCCG) and graded with the Clavien-Dindo (CD) classification
Readmission rate | 2014-2018
  Hospital readmissions during the 30 first days after hospital discharge
Length of stay | 2014-2018
  Postoperative stay from surgery to hospital discharge
Mortality rate | 2014-2018
  Mortality recorded during the 90 first days after surgery
Percentage of failure-to-rescue | 2014-2018
  Proportion of patients with a severe complication (Clavien-Dindo score >IIIa) dying during the first 90 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Javier Osorio, MD, PhD, Principal Investigator — Hospital Universitari de Bellvitge

IPD SHARING:
Plan to Share IPD: Yes
Report of global data description to all responsible surgeons of participant hospitals
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2020
Access Criteria: All responsible surgeons of participant hospitals

REFERENCES:
- [Background] Jerico C, Osorio J, Garcia-Erce JA, Pera M. Patient Blood Management strategies for iron deficiency anemia management in gastric cancer. Eur J Gastroenterol Hepatol. 2019 Apr;31(4):547-548. doi: 10.1097/MEG.0000000000001383. No abstract available. PMID 30829765
- [Background] Messager M, de Steur W, Boelens PG, Jensen LS, Mariette C, Reynolds JV, Osorio J, Pera M, Johansson J, Kolodziejczyk P, Roviello F, De Manzoni G, Monig SP, Allum WH; EURECCA Upper GI group (European Registration of Cancer Care). Description and analysis of clinical pathways for oesophago-gastric adenocarcinoma, in 10 European countries (the EURECCA upper gastro intestinal group - European Registration of Cancer Care). Eur J Surg Oncol. 2016 Sep;42(9):1432-47. doi: 10.1016/j.ejso.2016.01.001. Epub 2016 Feb 6. PMID 26898839
- [Background] Messager M, de Steur WO, van Sandick JW, Reynolds J, Pera M, Mariette C, Hardwick RH, Bastiaannet E, Boelens PG, van deVelde CJ, Allum WH; EURECCA Upper GI Group. Variations among 5 European countries for curative treatment of resectable oesophageal and gastric cancer: A survey from the EURECCA Upper GI Group (EUropean REgistration of Cancer CAre). Eur J Surg Oncol. 2016 Jan;42(1):116-22. doi: 10.1016/j.ejso.2015.09.017. Epub 2015 Sep 30. PMID 26461256
- [Background] Allum W, Osorio J. EURECCA oesophago-gastric cancer project. Cir Esp. 2016 May;94(5):255-6. doi: 10.1016/j.ciresp.2015.12.005. Epub 2016 Mar 2. No abstract available. English, Spanish. PMID 26944535
- [Result] Osorio J, Jerico C, Miranda C, Garsot E, Luna A, Miro M, Santamaria M, Artigau E, Rodriguez-Santiago J, Castro S, Feliu J, Aldeano A, Olona C, Momblan D, Ruiz D, Galofre G, Pros I, Garcia-Albeniz X, Lozano M, Pera M. Perioperative transfusion management in gastric cancer surgery: Analysis of the Spanish subset of the EURECCA oesophago-gastric cancer registry. Cir Esp (Engl Ed). 2018 Nov;96(9):546-554. doi: 10.1016/j.ciresp.2018.03.010. English, Spanish. PMID 29773261